CLINICAL TRIAL: NCT03635567
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Trial of Pembrolizumab (MK-3475) Plus Chemotherapy Versus Chemotherapy Plus Placebo for the First-Line Treatment of Persistent, Recurrent, or Metastatic Cervical Cancer (KEYNOTE-826)
Brief Title: Efficacy and Safety Study of First-line Treatment With Pembrolizumab (MK-3475) Plus Chemotherapy Versus Placebo Plus Chemotherapy in Women With Persistent, Recurrent, or Metastatic Cervical Cancer (MK-3475-826/KEYNOTE-826)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3475-826; MK-3475-826 (Other: MSD); KEYNOTE-826 (Other: MSD); 184183 (Registry Identifier: JAPAC-CTI); 2018-001440-53 (EudraCT Number)
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Uterine Cervical Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Paclitaxel; Cisplatin; Carboplatin; Bevacizumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab+Chemotherapy (Experimental): On Day 1 of each 21-day cycle, participants receive an intravenous (IV) infusion of pembrolizumab 200 mg for up to 35 cycles (up to approximately 2 years) PLUS Investigator choice of chemotherapy for up to 6 cycles (paclitaxel 175 mg/m^2 PLUS cisplatin 50 mg/m^2 WITH or WITHOUT bevacizumab 15 mg/kg per local label OR paclitaxel 175 mg/m^2 PLUS carboplatin Area Under the Curve (AUC) 5 for up to 6 cycles, WITH or WITHOUT bevacizumab 15 mg/kg per local label). All treatments are administered until disease progression or toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Paclitaxel; Drug: Cisplatin; Drug: Carboplatin; Biological: Bevacizumab
- Placebo+Chemotherapy (Placebo Comparator): On Day 1 of each 21-day cycle, participants receive an IV infusion of placebo (Normal Saline or Dextrose solution) for up to 35 cycles (up to approximately 2 years) PLUS Investigator choice of chemotherapy for up to 6 cycles (paclitaxel 175 mg/m^2 PLUS cisplatin 50 mg/m^2 WITH or WITHOUT bevacizumab 15 mg/kg per local label OR paclitaxel 175 mg/m^2 PLUS carboplatin AUC 5 for up to 6 cycles, WITH or WITHOUT bevacizumab 15 mg/kg per local label). All treatments are administered until disease progression or toxicity.
  Interventions: Drug: Paclitaxel; Drug: Cisplatin; Drug: Carboplatin; Biological: Bevacizumab; Drug: Placebo to pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab+Chemotherapy
Drug: Paclitaxel — IV infusion
  Other Names: TAXOL®
Drug: Cisplatin — IV infusion
  Other Names: PLATINOL®
Drug: Carboplatin — IV infusion
  Other Names: PARAPLATIN®
Biological: Bevacizumab — IV infusion
  Other Names: AVASTIN®
Drug: Placebo to pembrolizumab — IV infusion
  Other Names: Normal Saline or Dextrose solution
  Arms: Placebo+Chemotherapy

SUMMARY:
The purpose of this study is to assess the efficacy and safety of pembrolizumab (MK-3475) plus one of four platinum-based chemotherapy regimens compared to the efficacy and safety of placebo plus one of four platinum-based chemotherapy regimens in the treatment of adult women with persistent, recurrent, or metastatic cervical cancer. Possible chemotherapy regimens include: paclitaxel plus cisplatin with or without bevacizumab and paclitaxel plus carboplatin with or without bevacizumab.

The primary study hypotheses are that the combination of pembrolizumab plus chemotherapy is superior to placebo plus chemotherapy with respect to: 1) Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) as assessed by the Investigator, or, 2) Overall Survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Has persistent, recurrent, or metastatic squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix which has not been treated with systemic chemotherapy and is not amenable to curative treatment (such as with surgery and/or radiation). Prior chemotherapy utilized as a radiosensitizing agent and completed at least 2 weeks prior to randomization with resolution of all treatment-related toxicities is allowed. AEs due to previous treatments should be resolved to ≤ Grade 1 or baseline. Participants with ≤ Grade 2 neuropathy or ≤ Grade 2 alopecia are eligible.
* Not pregnant or breastfeeding, and at least one of the following conditions applies: a.) Not a woman of childbearing potential (WOCBP), b.) A WOCBP must agree to use effective contraception during the treatment period and for at least 120 days after the last dose of pembrolizumab/placebo and 210 days after the last dose of chemotherapy/bevacizumab
* Has measurable disease per RECIST 1.1 as assessed by the local site investigator/radiology
* Has provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated for prospective determination of Programmed Cell Death-Ligand 1 (PD-L1) status prior to randomization
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 within 14 days prior to randomization
* Has adequate organ function

Exclusion Criteria:

* A WOCBP who has a positive urine pregnancy test within 72 hours prior to randomization
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with known brain metastases may participate provided that the brain metastases have been previously treated (except with chemotherapy) and are radiographically stable.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, transitional cell carcinoma of urothelial cancer, or carcinoma in situ (e.g. breast cancer) that have undergone potentially curative therapy are not excluded.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in doses exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to randomization
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of Hepatitis B or known active Hepatitis C virus infection
* Has a known history of active tuberculosis (TB; Bacillus tuberculosis)
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX 40, CD137)
* Has received prior systemic chemotherapy for treatment of cervical cancer.
* Has not recovered adequately from toxicity and/or complications from major surgery prior to randomization
* Has received prior radiotherapy within 2 weeks prior to randomization. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
* Has received a live vaccine within 30 days prior to randomization
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has a contraindication or hypersensitivity to any component of cisplatin, carboplatin, paclitaxel, or bevacizumab
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to randomization
* Is pregnant or breastfeeding or expecting to conceive within the projected duration of the study, starting with the screening visit through 120 days following last dose of pembrolizumab/placebo and 210 days following last dose of chemotherapy/bevacizumab
* Has had an allogeneic tissue/solid organ transplant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 617 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2024-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (149):
- United States (20):
  - Alaska Women's Cancer Care ( Site 1770), Anchorage, Alaska
  - Arizona Oncology Associates, PC- HAL ( Site 8005), Phoenix, Arizona
  - UC Irvine Health ( Site 1796), Orange, California
  - Smilow Cancer Hospital at Yale New Haven ( Site 1809), New Haven, Connecticut
  - H. Lee Moffitt Cancer Center and Research Institute ( Site 1754), Tampa, Florida
  - Georgia Cancer Center at Augusta University ( Site 1767), Augusta, Georgia
  - Barbara Ann Karmanos Cancer Institute ( Site 1785), Detroit, Michigan
  - Henry Ford Health System ( Site 1810), Detroit, Michigan
  - Washington University School of Medicine ( Site 1779), St Louis, Missouri
  - Cancer Institute of New Jersey at University Hospital ( Site 1762), Newark, New Jersey
  - Holy Name Medical Center ( Site 1776), Teaneck, New Jersey
  - Mount Sinai Chelsea ( Site 1760), New York, New York
  - Columbia University Medical Center ( Site 1800), New York, New York
  - OSU Wexner Medical Center ( Site 1817), Hilliard, Ohio
  - University of Oklahoma- Stephenson Oklahoma Cancer Center ( Site 1784), Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute, LLC ( Site 1768), Tulsa, Oklahoma
  - MUSC Hollings Cancer Center ( Site 1819), Charleston, South Carolina
  - West Cancer Center - East Campus ( Site 1763), Germantown, Tennessee
  - Texas Oncology-San Antonio Medical Center ( Site 8001), San Antonio, Texas
  - Seattle Cancer Care Alliance ( Site 1777), Seattle, Washington
- Argentina (6):
  - Centro de Oncologia e Investigacion Buenos Aires COIBA ( Site 1006), Berazategui, Buenos Aires
  - Hospital Aleman ( Site 1005), Buenos Aires
  - Hospital de Oncologia Angel Roffo ( Site 1003), Buenos Aires
  - Instituto Medico Especializado Alexander Fleming ( Site 1009), Buenos Aires
  - Centro Oncologico Riojano Integral ( Site 1004), La Rioja
  - Centro Medico San Roque ( Site 1001), San Miguel de Tucumán
- Australia (5):
  - Royal North Shore Hospital ( Site 1514), St Leonards, New South Wales
  - Mater Misericordiae Ltd Mater Cancer Care Centre ( Site 1521), South Brisbane, Queensland
  - Flinders Medical Centre ( Site 1513), Bedford Park, South Australia
  - St John of God Subiaco Hospital ( Site 1512), Subiaco, Western Australia
  - Monash Health-Monash Medical Centre ( Site 1519), Clayton
- Canada (15):
  - Tom Baker Cancer Centre ( Site 1728), Calgary, Alberta
  - BC Cancer-Kelowna - Sindi Ahluwalia Hawkins Centre ( Site 1734), Kelowna, British Columbia
  - BC Cancer - Vancouver Center ( Site 1722), Vancouver, British Columbia
  - CancerCare Manitoba ( Site 1725), Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre ( Site 1731), Halifax, Nova Scotia
  - Juravinski Cancer Centre ( Site 1735), Hamilton, Ontario
  - London Regional Cancer Program - London HSC ( Site 1723), London, Ontario
  - The Ottawa Hospital Cancer Centre ( Site 1736), Ottawa, Ontario
  - Sunnybrook Research Institute ( Site 1733), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 1732), Toronto, Ontario
  - CIUSSS du Saguenay-Lac-St-Jean ( Site 1729), Chicoutimi, Quebec
  - CIUSSS de l Est de L Ile de Montreal - Hopital Maisonneuve-Rosemont ( Site 1726), Montreal, Quebec
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 1721), Montreal, Quebec
  - CHU de Quebec-Universite Laval-Hotel Dieu de Quebec ( Site 1724), Québec, Quebec
  - CIUSSS de l Estrie - CHUS - Centre Hosp. Univ. Sherbrooke ( Site 1730), Sherbrooke, Quebec
- Chile (5):
  - Oncocentro ( Site 1065), Viña del Mar, Región de Valparaíso
  - Fundacion Arturo Lopez Perez FALP ( Site 1061), Santiago
  - Sociedad Oncovida S.A. ( Site 1069), Santiago
  - Centro de Cancer Nuestra Senora de la Esperanza ( Site 1063), Santiago
  - Instituto Clinico Oncologico del Sur ( Site 1062), Temuco
- Colombia (6):
  - Sociedad de Oncologia y Hematologia del Cesar Ltda. ( Site 1103), Valledupar, Cesar Department
  - Instituto Nacional de Cancerologia E.S.E ( Site 1095), Bogota, Cundinamarca
  - Hemato Oncologos S.A. ( Site 1100), Cali, Valle del Cauca Department
  - Biomelab S A S ( Site 1104), Barranquilla
  - Oncomedica S.A. ( Site 1098), Montería
  - Instituto Cancerologico de Narino Ltda ( Site 1097), Pasto
- France (5):
  - Centre Jean Perrin ( Site 1181), Clermont-Ferrand
  - Institut Paoli Calmettes ( Site 1182), Marseille
  - Groupe Hospitalier Broca Cochin Hotel Dieu ( Site 1183), Paris
  - Centre Eugene Marquis ( Site 1187), Rennes
  - Institut Curie - Centre Rene Huguenin ( Site 1185), Saint-Cloud
- Germany (9):
  - Universitaetsklinikum Carl Gustav Carus ( Site 1211), Dresden
  - Universitaetsklinikum Duesseldorf ( Site 1220), Düsseldorf
  - Universitatsklinikum Essen AoR ( Site 1213), Essen
  - Universitatsklinikum Hamburg-Eppendorf ( Site 1212), Hamburg
  - Gynoncological Practice Lueck. Schrader. Noeding ( Site 1224), Hanover
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel ( Site 1214), Kiel
  - Rotkreuzklinikum Muenchen gGmbH. Studienzentrale Frauenklinik ( Site 1225), München
  - Klinikum Oldenburg AoeR ( Site 1218), Oldenburg
  - Universitaet Regensburg ( Site 1221), Regensburg
- Israel (7):
  - Soroka Medical Center ( Site 1363), Beersheba
  - Rambam Medical Center ( Site 1364), Haifa
  - Shaare Zedek Medical Center ( Site 1366), Jerusalem
  - Hadassah Medical Center. Ein Kerem ( Site 1367), Jerusalem
  - Rabin Medical Center ( Site 1365), Petah Tikva
  - Chaim Sheba Medical Center ( Site 1361), Ramat Gan
  - Sourasky Medical Center ( Site 1362), Tel Aviv
- Italy (6):
  - Centro di Riferimento Oncologico de Aviano Istituto Nazionale Tumori ( Site 1243), Aviano
  - A.O. Universitaria Policlinico S. Orsola-Malpighi ( Site 1245), Bolgna
  - Istituto Nazionale Tumori ( Site 1251), Milan
  - Istituto Europeo di Oncologia ( Site 1250), Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 1242), Napoli
  - Policlinico Universitario -Agostino Gemelli ( Site 1241), Roma
- Japan (14):
  - The Jikei University Kashiwa Hospital ( Site 1701), Kashiwa, Chiba
  - National Cancer Center Hospital East ( Site 1704), Kashiwa, Chiba
  - Ehime University Hospital ( Site 1693), Tōon, Ehime
  - Kurume University Hospital ( Site 1692), Kurume, Fukuoka
  - National Hospital Organization Hokkaido Cancer Center ( Site 1700), Sapporo, Hokkaido
  - Hyogo Cancer Center ( Site 1705), Akashi, Hyōgo
  - Iwate Medical University Hospital ( Site 1695), Shiwa-gun, Iwate
  - University of the Ryukyus Hospital ( Site 1706), Nakagami-gun, Okinawa
  - Saitama Medical University International Medical Center ( Site 1691), Hidaka, Saitama
  - Shizuoka Cancer Center Hospital and Research Institute ( Site 1703), Sunto-gun, Shizuoka
  - National Cancer Center Hospital ( Site 1702), Tokyo
  - The Jikei University Hospital ( Site 1697), Tokyo
  - The Cancer Institute Hospital of JFCR ( Site 1698), Tokyo
  - Keio University Hospital ( Site 1699), Tokyo
- Mexico (7):
  - Medical Care and Research S.A. de C.V. ( Site 1135), Mérida, Yucatán
  - Centro Estatal de Cancerologia de Chihuahua ( Site 1123), Chihuahua City
  - Consultorio de Medicina Especializada del Sector Privado ( Site 1129), Mexico City
  - CRYPTEX Investigacion Clinica S.A. de C.V. ( Site 1127), Mexico City
  - Instituto Nacional de Cancerologia. ( Site 1130), México
  - Centro de Urologia Avanzada del Noreste S.A. de C.V. ( Site 1125), San Pedro Garza García
  - Faicic S de RL de CV ( Site 1133), Veracruz
- Peru (7):
  - Hospital de Alta Complejidad de La Libertad Virgen de La Puerta ( Site 1152), Trujillo, La Libertad
  - Centro Medico Monte Carmelo ( Site 1156), Arequipa
  - Hospital Nacional Guillermo Almenara Irigoyen ( Site 1158), Lima
  - Instituto de Oncologia y Radioterapia Clinica Ricardo Palma ( Site 1157), Lima
  - Instituto Nacional de Enfermedades Neoplasicas ( Site 1153), Lima
  - Hospital Nacional Arzobispo Loayza ( Site 1159), Lima
  - Hospital Nacional Maria Auxiliadora ( Site 1155), Lima
- Russia (9):
  - Republican Clinical Oncology Dispensary of Tatarstan MoH ( Site 1331), Kazan'
  - FSBI National Medical Oncology Research Center n.a. N.N. Blokhina ( Site 1334), Moscow
  - Medical Rehabilitation Center ( Site 1337), Moscow
  - Novosibirsk Regional Clinical Oncology Dispensary ( Site 1358), Novosibirsk
  - National Medical Research Center of Oncology n.a. N. N. Petrov ( Site 1348), Saint Petersburg
  - Municipal Clinical Oncology Center ( Site 1346), Saint Petersburg
  - National Research Ogarev Mordovia State University ( Site 1347), Saransk
  - Tomsk Scientific Research Institute of Oncology ( Site 1360), Tomsk
  - Republican Clinical Oncology Dispensary of Republic of Bashkortostan ( Site 1345), Ufa
- South Korea (4):
  - Keimyung University Dongsan Medical Center ( Site 1603), Daegu
  - Seoul National University Hospital ( Site 1602), Seoul
  - Asan Medical Center ( Site 1601), Seoul
  - Samsung Medical Center ( Site 1604), Seoul
- Spain (5):
  - Onkologikoa - Instituto Oncologico de San Sebastian ( Site 1275), Doniostia - San Sebastian, Guipuzcoa
  - Hospital Quiron Madrid ( Site 1277), Pozuelo de Alarcón, Madrid
  - Hospital Germans Trias i Pujol. ICO de Badalona ( Site 1276), Badalona
  - MD Anderson Cancer Center Madrid ( Site 1273), Madrid
  - Hospital Universitario Virgen Macarena ( Site 1274), Seville
- Taiwan (6):
  - Kaohsiung Veterans General Hospital ( Site 1632), Kaohsiung City
  - China Medical University Hospital ( Site 1635), Taichung
  - Taichung Veterans General Hospital ( Site 1634), Taichung
  - Koo Foundation Sun Yat-Sen Cancer Center ( Site 1636), Taipei
  - Taipei Veterans General Hospital ( Site 1631), Taipei
  - Chang Gung Medical Foundation. Linkou ( Site 1633), Taoyuan District
- Turkey (Türkiye) (7):
  - Baskent Adana Dr Turgut Noyan Uygulama ve Arastirma Merkezi ( Site 1457), Adana
  - Hacettepe University Medical Faculty ( Site 1459), Ankara
  - Baskent Universitesi Ankara Hastanesi ( Site 1451), Ankara
  - Akdeniz Universitesi Tip Fakultesi ( Site 1453), Antalya
  - Medeniyet University Goztepe Egitim ve Arastırma Hast. Merdivenkoy ( Site 1458), Istanbul
  - Ege University Medical Faculty Tulay Aktas Oncology Hospital ( Site 1456), Izmir
  - Necmettin Erbakan Universitesi Meram Tip Fakultesi Hastanesi ( Site 1452), Konya
- Ukraine (6):
  - City Clinical Hosp.4 of DCC ( Site 1482), Dnipropetrovsk
  - MI Precarpathian Clinical Oncology Center ( Site 1487), Ivano-Frankivsk
  - Communal non profit enterprise Regional Clinical Oncology Center ( Site 1489), Kharkiv
  - National Cancer Institute of the MoH of Ukraine ( Site 1484), Kyiv
  - MI Odessa Regional Oncological Centre ( Site 1493), Odesa
  - Medical Centre LLC Oncolife ( Site 1485), Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Monk BJ, Colombo N, Tewari KS, Dubot C, Caceres MV, Hasegawa K, Shapira-Frommer R, Salman P, Yanez E, Gumus M, Olivera Hurtado de Mendoza M, Samouelian V, Castonguay V, Arkhipov A, Tekin C, Li K, Keefe SM, Lorusso D; KEYNOTE-826 Investigators. First-Line Pembrolizumab + Chemotherapy Versus Placebo + Chemotherapy for Persistent, Recurrent, or Metastatic Cervical Cancer: Final Overall Survival Results of KEYNOTE-826. J Clin Oncol. 2023 Dec 20;41(36):5505-5511. doi: 10.1200/JCO.23.00914. Epub 2023 Nov 1. PMID 37910822
- [Derived] Kim YM, Nishio S, Kim SI, Hasegawa K, Dubot C, Caceres MV, Tewari KS, Lorusso D, Lee JW, Liou WS, Li K, Tekin C, Colombo N, Monk BJ. Pembrolizumab plus chemotherapy with or without bevacizumab in East Asian participants with persistent, recurrent, or metastatic cervical cancer: results from KEYNOTE-826 final analysis. J Gynecol Oncol. 2025 Jul;36(4):e110. doi: 10.3802/jgo.2025.36.e110. PMID 40590325
- [Derived] Monk BJ, van Mens S, Hale O, Boer J, van Hees F, Swami S, Muston D, Tekin C, Keefe S, Monberg M. Cost-Effectiveness of Pembrolizumab as First-Line Treatment in Patients with Persistent, Recurrent, or Metastatic Cervical Cancer in the United States. Oncol Ther. 2025 Mar;13(1):85-98. doi: 10.1007/s40487-024-00311-5. Epub 2024 Nov 5. PMID 39499492
- [Derived] Tewari KS, Colombo N, Monk BJ, Dubot C, Caceres MV, Hasegawa K, Shapira-Frommer R, Salman P, Yanez E, Gumus M, Olivera Hurtado de Mendoza M, Samouelian V, Castonguay V, Arkhipov A, Tekin C, Li K, Toker S, Keefe SM, Lorusso D. Pembrolizumab or Placebo Plus Chemotherapy With or Without Bevacizumab for Persistent, Recurrent, or Metastatic Cervical Cancer: Subgroup Analyses From the KEYNOTE-826 Randomized Clinical Trial. JAMA Oncol. 2024 Feb 1;10(2):185-192. doi: 10.1001/jamaoncol.2023.5410. PMID 38095881
- [Derived] Monk BJ, Tewari KS, Dubot C, Caceres MV, Hasegawa K, Shapira-Frommer R, Salman P, Yanez E, Gumus M, Hurtado de Mendoza MO, Samouelian V, Castonguay V, Arkhipov A, Tekin C, Li K, Martin Nguyen A, Monberg MJ, Colombo N, Lorusso D. Health-related quality of life with pembrolizumab or placebo plus chemotherapy with or without bevacizumab for persistent, recurrent, or metastatic cervical cancer (KEYNOTE-826): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2023 Apr;24(4):392-402. doi: 10.1016/S1470-2045(23)00052-9. Epub 2023 Mar 3. PMID 36878237
- [Derived] Colombo N, Dubot C, Lorusso D, Caceres MV, Hasegawa K, Shapira-Frommer R, Tewari KS, Salman P, Hoyos Usta E, Yanez E, Gumus M, Olivera Hurtado de Mendoza M, Samouelian V, Castonguay V, Arkhipov A, Toker S, Li K, Keefe SM, Monk BJ; KEYNOTE-826 Investigators. Pembrolizumab for Persistent, Recurrent, or Metastatic Cervical Cancer. N Engl J Med. 2021 Nov 11;385(20):1856-1867. doi: 10.1056/NEJMoa2112435. Epub 2021 Sep 18. PMID 34534429
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26852&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 883 participants were screened and 617 participants were randomized to receive either Pembrolizumab+Chemotherapy or Placebo+Chemotherapy.
Groups:
- Pembrolizumab+Chemotherapy: On Day 1 of each 21-day cycle, participants received an intravenous (IV) infusion of pembrolizumab 200 mg for up to 35 cycles (up to approximately 2 years) PLUS Investigator choice of chemotherapy for up to 6 cycles (paclitaxel 175 mg/m^2 PLUS cisplatin 50 mg/m^2 WITH or WITHOUT bevacizumab 15 mg/kg per local label OR paclitaxel 175 mg/m^2 PLUS carboplatin Area Under the Curve (AUC) 5 for up to 6 cycles, WITH or WITHOUT bevacizumab 15 mg/kg per local label). All treatments were administered until disease progression or toxicity. Eligible participants who stopped the initial course of pembrolizumab with Stable Disease (SD) or better but progressed after discontinuation may have been able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
- Placebo+Chemotherapy: On Day 1 of each 21-day cycle, participants received an IV infusion of placebo (Normal Saline or Dextrose solution) for up to 35 cycles (up to approximately 2 years) PLUS Investigator choice of chemotherapy for up to 6 cycles (paclitaxel 175 mg/m^2 PLUS cisplatin 50 mg/m^2 WITH or WITHOUT bevacizumab 15 mg/kg per local label OR paclitaxel 175 mg/m^2 PLUS carboplatin AUC 5 for up to 6 cycles, WITH or WITHOUT bevacizumab 15 mg/kg per local label). All treatments were administered until disease progression or toxicity.
Period: Overall Study
Arm/Group | Pembrolizumab+Chemotherapy | Placebo+Chemotherapy
Started | 308 | 309
Treated | 307 | 309
Received Second Course of Pembrolizumab | 12 | 0
Completed | 0 | 0
Not Completed | 308 | 309
Not completed — Lost to Follow-up | 4 | 1
Not completed — Withdrawal by Subject | 11 | 16
Not completed — Sponsor Decision | 99 | 57
Not completed — Death | 194 | 235

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab+Chemotherapy | Placebo+Chemotherapy | Total
Number analyzed (Participants) | 308 | 309 | 617
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.7 (11.9) | 50.7 (12.7) | 51.2 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 308 | 309 | 617
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 109 | 121 | 230
  Not Hispanic or Latino | 193 | 184 | 377
  Unknown or Not Reported | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 18 | 21 | 39
  Asian | 65 | 45 | 110
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 170 | 190 | 360
  More than one race | 32 | 34 | 66
  Unknown or Not Reported | 19 | 17 | 36
Programmed Cell Death-Ligand 1 (PD-L1) Combined Positive Score (CPS) Status [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression level by immunohistochemistry assay using tumor tissue. Randomization of participants in the study were stratified by their PD-L1 CPS at baseline (PD-L1 CPS<1, 1≤ PD-L1 CPS<10, or PD-L1 CPS≥10).
  Participants
    PD-L1 CPS<1 | 35 | 34 | 69
    1≤ PD-L1 CPS<10 | 115 | 116 | 231
    PD-L1 CPS≥10 | 158 | 159 | 317
Metastatic at Initial Diagnosis [Count of Participants; unit: Participants] — Randomization of participants was stratified by whether they were metastatic at initial diagnosis (Yes or No). Metastatic was defined as Stage IVB based on the Fédération Internationale de Gynécologie et d'Obstétrique (FIGO) (2009).
  Participants
    Yes | 94 | 96 | 190
    No | 214 | 213 | 427
Investigator Choice to Use Bevacizumab [Count of Participants; unit: Participants] — Randomization of participants was stratified by the Investigator's choice for the participant to receive bevacizumab (Yes or No).
  Participants
    Yes | 196 | 193 | 389
    No | 112 | 116 | 228

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Investigator in Participants With Programmed Cell Death-Ligand 1 (PD-L1) Combined Positive Score (CPS) ≥1
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as ≥ 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. The PFS per RECIST 1.1 as assessed by Investigator for all randomized participants with PD-L1 CPS ≥1 is presented.
Time Frame: Up to approximately 46 months
Population: All randomized participants with PD-L1 CPS ≥1 based on the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Chemotherapy | Placebo+Chemotherapy
Number analyzed (Participants) | 273 | 275
Months | 10.5 [9.7 to 12.3] | 8.2 [6.3 to 8.5]
Statistical Analysis 1: Comparison: Pembrolizumab+Chemotherapy vs Placebo+Chemotherapy; Treatment comparison (hazard ratio [HR]) was based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by metastatic at initial diagnosis (FIGO [2009] stage IVB) (yes or no), bevacizumab use (yes or no), and PD-L1 status (CPS<1, CPS 1 to <10, or CPS ≥10); Test type: Other; p < 0.0001, Stratified Log-Rank — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Nominal p-value based on log-rank test stratified by metastatic at initial diagnosis (FIGO [2009] stage IVB), bevacizumab use, and PD-L1 status; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.47 to 0.71]

2. Primary Outcome: PFS Per RECIST 1.1 as Assessed by Investigator in All Participants
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as ≥ 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. The PFS per RECIST 1.1 as assessed by Investigator for all randomized participants is presented.
Time Frame: Up to approximately 46 months
Population: All randomized participants based on the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Chemotherapy | Placebo+Chemotherapy
Number analyzed (Participants) | 308 | 309
Months | 10.4 [9.1 to 12.2] | 8.2 [6.4 to 8.4]
Statistical Analysis 1: Comparison: Pembrolizumab+Chemotherapy vs Placebo+Chemotherapy; Treatment comparison (HR) was based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by metastatic at initial diagnosis (FIGO [2009] stage IVB) (yes or no), bevacizumab use (yes or no), and PD-L1 status (CPS<1, CPS 1 to <10, or CPS ≥10); Test type: Other; p < 0.0001, Stratified Log-Rank — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.50 to 0.74]

3. Primary Outcome: PFS Per RECIST 1.1 as Assessed by Investigator in Participants With PD-L1 CPS ≥10
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as ≥ 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. The PFS per RECIST 1.1 as assessed by Investigator for all randomized participants with PD-L1 CPS ≥10 is presented.
Time Frame: Up to approximately 46 months
Population: All randomized participants with PD-L1 CPS ≥10 based on the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Chemotherapy | Placebo+Chemotherapy
Number analyzed (Participants) | 158 | 159
Months | 10.4 [8.9 to 15.1] | 8.1 [6.2 to 8.8]
Statistical Analysis 1: Comparison: Pembrolizumab+Chemotherapy vs Placebo+Chemotherapy; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.0001, Stratified Log-Rank — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.40 to 0.68]

4. Primary Outcome: Overall Survival (OS) in Participants With PD-L1 CPS ≥1
Description: OS was defined as the time from randomization to death due to any cause. The OS for all randomized participants with PD-L1 CPS ≥1 is presented.
Time Frame: Up to approximately 46 months
Population: All randomized participants with PD-L1 CPS ≥1 based on the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Chemotherapy | Placebo+Chemotherapy
Number analyzed (Participants) | 273 | 275
Months | 28.6 [22.1 to 38.0] | 16.5 [14.5 to 20.0]
Statistical Analysis 1: Comparison: Pembrolizumab+Chemotherapy vs Placebo+Chemotherapy; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.0001, Stratified Log-Rank — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.49 to 0.74]

5. Primary Outcome: OS in All Participants
Description: OS was defined as the time from randomization to death due to any cause. The OS for all randomized participants is presented.
Time Frame: Up to approximately 46 months
Population: All randomized participants based on the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Chemotherapy | Placebo+Chemotherapy
Number analyzed (Participants) | 308 | 309
Months | 26.4 [21.3 to 32.5] | 16.8 [14.6 to 19.4]
Statistical Analysis 1: Comparison: Pembrolizumab+Chemotherapy vs Placebo+Chemotherapy; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.0001, Stratified Log-Rank — No formal hypothesis testing performed; nominal p-value based on log-rank test provided for treatment comparison; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.52 to 0.77]

6. Primary Outcome: OS in Participants With PD-L1 CPS ≥10
Description: OS was defined as the time from randomization to death due to any cause. The OS for all randomized participants with PD-L1 CPS ≥10 is presented.
Time Frame: Up to approximately 46 months
Population: All randomized participants with PD-L1 CPS ≥10 based on the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Chemotherapy | Placebo+Chemotherapy
Number analyzed (Participants) | 158 | 159
Months | 29.6 [20.6 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 17.4 [14.0 to 24.7]
Statistical Analysis 1: Comparison: Pembrolizumab+Chemotherapy vs Placebo+Chemotherapy; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.0001, Stratified Log-Rank — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.44 to 0.78]

7. Secondary Outcome: Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by Investigator
Description: ORR was defined as the percentage of the participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters). The ORR per RECIST 1.1 as assessed by Investigator is presented.
Time Frame: Up to approximately 46 months
Population: All randomized participants based on the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab+Chemotherapy | Placebo+Chemotherapy
Number analyzed (Participants) | 308 | 309
Percentage of Participants | 66.2 [60.7 to 71.5] | 51.5 [45.7 to 57.2]
Statistical Analysis 1: Comparison: Pembrolizumab+Chemotherapy vs Placebo+Chemotherapy; Treatment comparison was based on Miettinen & Nurminen method stratified by metastatic at initial diagnosis (FIGO [2009] stage IVB) (yes or no), bevacizumab use (yes or no), and PD-L1 status (CPS<1, CPS 1 to <10, or CPS ≥10); Test type: Other; p = 0.0001, Miettinen & Nurminen method — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Difference in Percentage = 14.9, 95% CI 2-sided [7.4 to 22.3]

8. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 as Assessed by Investigator
Description: For participants who demonstrate CR or PR, DOR was defined as the time from first documented evidence of CR or PR until disease progression or death. The DOR per RECIST 1.1 as assessed by Investigator is presented.
Time Frame: Up to approximately 46 months
Population: All randomized participants based on the treatment group to which they were randomized who demonstrated CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Chemotherapy | Placebo+Chemotherapy
Number analyzed (Participants) | 204 | 159
Months | 18.0 [10.5 to 32.3] | 10.4 [8.3 to 13.3]

9. Secondary Outcome: Percentage of Participants That Were PFS Event-Free (PFS Rate) at Month 12 Per RECIST 1.1 as Assessed by Investigator
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as ≥ 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. PFS Rate was defined as the percentage of participants that were PFS event-free at Month 12. The PFS Rate per RECIST 1.1 as assessed by Investigator at Month 12 is presented.
Time Frame: 12 months
Population: All randomized participants based on the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab+Chemotherapy | Placebo+Chemotherapy
Number analyzed (Participants) | 308 | 309
Percentage of Participants | 44.7 [38.9 to 50.4] | 33.1 [27.7 to 38.7]

10. Secondary Outcome: PFS Per RECIST 1.1 as Assessed by Blinded Independent Central Review (BICR)
Description: PFS was defined as the time from randomization to the first documented PD or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as ≥ 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. The PFS per RECIST 1.1 as assessed by BICR is presented.
Time Frame: Up to approximately 46 months
Population: All randomized participants based on the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Chemotherapy | Placebo+Chemotherapy
Number analyzed (Participants) | 308 | 309
Months | 12.3 [10.3 to 17.9] | 8.3 [8.1 to 9.0]
Statistical Analysis 1: Comparison: Pembrolizumab+Chemotherapy vs Placebo+Chemotherapy; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.0001, Stratified Log-Rank — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.49 to 0.74]

11. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experienced an AE is presented.
Time Frame: Up to approximately 66 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Number of participants
Arm/Group | Pembrolizumab+Chemotherapy | Placebo+Chemotherapy
Number analyzed (Participants) | 307 | 309
Number of participants | 305 | 307

12. Secondary Outcome: Number of Participants Who Experienced a Serious AE (SAE)
Description: An SAE was defined as any untoward medical occurrence that, at any dose: a.) Resulted in death; b.) Was life-threatening; c.) Required inpatient hospitalization or prolongation of existing hospitalization; d.) Resulted in persistent or significant disability/incapacity; e.) Was a congenital anomaly/birth defect; f.) Other important medical events; h.) Was a new cancer (that is not a condition of the study) or i.) Was associated with an overdose. The number of participants who experienced an SAE is presented.
Time Frame: Up to approximately 66 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Number of Participants
Arm/Group | Pembrolizumab+Chemotherapy | Placebo+Chemotherapy
Number analyzed (Participants) | 307 | 309
Number of Participants | 157 | 132

13. Secondary Outcome: Number of Participants Who Experienced an Immune-related AE (irAE)
Description: AEs associated with pembrolizumab exposure may be a result of an immune response. These irAEs may occur shortly after the first dose or several months after the last dose of pembrolizumab treatment and may affect more than one body system simultaneously. For this study irAEs included, but were not limited to: -Pneumonitis;
  * Diarrhea/Colitis;
  * Aspartate transaminase (AST)/Alanine transaminase (ALT) elevation or Increased bilirubin;
  * Type 1 diabetes mellitus or Hyperglycemia;
  * Hypophysitis;
  * Hyperthyroidism;
  * Hypothyroidism;
  * Nephritis and Renal dysfunction; and
  * Myocarditis. The number of participants who experienced an irAE is presented.
Time Frame: Up to approximately 66 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Number of Participants
Arm/Group | Pembrolizumab+Chemotherapy | Placebo+Chemotherapy
Number analyzed (Participants) | 307 | 309
Number of Participants | 134 | 92

14. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 63 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Number of Participants
Arm/Group | Pembrolizumab+Chemotherapy | Placebo+Chemotherapy
Number analyzed (Participants) | 307 | 309
Number of Participants | 126 | 92

15. Secondary Outcome: Number of Participants With a 10-point Change From Baseline in Quality of Life (QoL) Based on the European Organisation for the Research & Treatment of Cancer (EORTC) QoL Questionnaire-30 (QLQ-C30) Combined Global Score
Description: The EORTC QLQ-C30 is a questionnaire to assess the quality of life of cancer patients. Participant responses to "How would you rate your overall health during the past week?" (Item 29) and "How would you rate your overall quality of life during the past week?" (Item 30) are scored on a 7-point scale (1= Very poor to 7=Excellent). Raw scores are standardized with linear transformation so that scores range from 0-100. A higher combined score indicates a better overall health status. Participant post-baseline scores were classified based on change from baseline, "Improved": a ≥10-point improvement in score and confirmed by the next visit; "Stable": a ≥10-point increase or <10-point change in score OR a <10-point change in score and a ≥10-point increase in score at the next visit; or "Deteriorated": a ≥10-point deterioration in score when the criteria for improvement/stability weren't met. Participants who didn't meet "Improved", "Stable", or "Deteriorated" criteria reported as "Other".
Time Frame: Baseline (Cycle 1 Day 1: Predose) and up to approximately 46 months
Population: Per protocol, all randomized participants who received at least one dose of study treatment and completed at least one EORTC QLQ-C30 assessment were analyzed. Participants with no EORTC QLQ-C30 assessment were not included in the analysis.
Measure: Number; unit: Number of Participants
Arm/Group | Pembrolizumab+Chemotherapy | Placebo+Chemotherapy
Number analyzed (Participants) | 279 | 282
Number of Participants
  Improved | 122 | 86
  Stable | 106 | 139
  Deteriorated | 42 | 48
  Other | 9 | 9

ADVERSE EVENTS:
Time Frame: Up to approximately 66 months
Description: Serious and Other adverse events (AEs) included all participants who received ≥1 dose of study drug. All-Cause Mortality included all randomized participants. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs. Data are reported by treatment received.
Groups:
- Pembrolizumab (Second Course): Eligible participants received up to 17 additional administrations (up to approximately 1 year) of pembrolizumab 200 mg IV on Day 1 of each 21-day cycle.
Arm/Group | Pembrolizumab+Chemotherapy | Placebo+Chemotherapy | Pembrolizumab (Second Course)
All-Cause Mortality (participants affected / at risk) | 195/308 | 241/309 | 4/12
Serious Adverse Events (participants affected / at risk) | 157/307 | 132/309 | 4/12
Other Adverse Events (participants affected / at risk) | 298/307 | 299/309 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab+Chemotherapy (N=307) | Placebo+Chemotherapy (N=309) | Pembrolizumab (Second Course) (N=12)
Anaemia (Blood and lymphatic system disorders) | 14 (14) | 12 (14) | 0 (0)
Bicytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 21 (25) | 13 (14) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (5) | 3 (3) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (3) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 1 (1) | 0 (0)
Bundle branch block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 3 (3) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Optic neuropathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 2 (2) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (4) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Rectal perforation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 3 (3) | 3 (3) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0)
Medical device site laceration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pseudocyst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 9 (9) | 5 (5) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (2) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 3 (3) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 2 (2) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute hepatitis B (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Cellulitis (Infections and infestations) | 1 (2) | 2 (2) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fournier's gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster meningoradiculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected fistula (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infected lymphocele (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pelvic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 7 (7) | 0 (0)
Psoas abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 4 (4) | 2 (4) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Pyometra (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 8 (8) | 5 (5) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 16 (17) | 20 (23) | 1 (2)
Urosepsis (Infections and infestations) | 2 (2) | 4 (5) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural urine leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radiation proctitis (Injury, poisoning and procedural complications) | 4 (6) | 2 (2) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Autoimmune myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ovarian cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalitis autoimmune (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Idiopathic intracranial hypertension (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 2 (2) | 2 (2) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Stent malfunction (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 11 (13) | 5 (6) | 0 (0)
Bladder diverticulum (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 5 (6) | 4 (4) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 4 (4) | 4 (4) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Postrenal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 3 (3) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urethral fistula (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 3 (3) | 0 (0)
Urinoma (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urogenital fistula (Renal and urinary disorders) | 5 (5) | 2 (2) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 8 (8) | 10 (10) | 1 (1)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 0 (0)
Vaginal fistula (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 5 (5) | 4 (5) | 0 (0)
Vulval ulceration (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 2 (2) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 3 (3) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vena cava embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab+Chemotherapy (N=307) | Placebo+Chemotherapy (N=309) | Pembrolizumab (Second Course) (N=12)
Anaemia (Blood and lymphatic system disorders) | 182 (264) | 159 (247) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 40 (71) | 33 (55) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 15 (29) | 7 (7) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 71 (142) | 58 (115) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 60 (90) | 60 (101) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 24 (26) | 9 (10) | 0 (0)
Hypothyroidism (Endocrine disorders) | 59 (65) | 31 (33) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 50 (66) | 52 (78) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 16 (18) | 12 (13) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 30 (43) | 30 (41) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 10 (11) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 89 (143) | 101 (147) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 111 (203) | 93 (174) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 20 (24) | 15 (19) | 1 (2)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 (11) | 13 (14) | 1 (1)
Nausea (Gastrointestinal disorders) | 122 (265) | 135 (287) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 16 (26) | 15 (20) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 22 (26) | 22 (30) | 1 (1)
Vomiting (Gastrointestinal disorders) | 81 (127) | 85 (142) | 1 (1)
Asthenia (General disorders) | 64 (122) | 66 (128) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 88 (148) | 85 (150) | 0 (0)
Mucosal inflammation (General disorders) | 23 (32) | 10 (14) | 0 (0)
Oedema peripheral (General disorders) | 32 (38) | 30 (36) | 0 (0)
Pyrexia (General disorders) | 51 (78) | 44 (61) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 13 (14) | 1 (1)
Nasopharyngitis (Infections and infestations) | 20 (26) | 11 (13) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 13 (19) | 16 (21) | 0 (0)
Urinary tract infection (Infections and infestations) | 67 (123) | 74 (111) | 0 (0)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 8 (8) | 3 (3) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 17 (24) | 12 (17) | 0 (0)
Alanine aminotransferase increased (Investigations) | 45 (67) | 29 (37) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 35 (57) | 24 (32) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 27 (33) | 18 (20) | 1 (1)
Blood creatinine increased (Investigations) | 28 (44) | 34 (42) | 0 (0)
Neutrophil count decreased (Investigations) | 56 (152) | 48 (143) | 0 (0)
Platelet count decreased (Investigations) | 49 (99) | 42 (69) | 1 (1)
Weight decreased (Investigations) | 35 (35) | 37 (38) | 0 (0)
White blood cell count decreased (Investigations) | 37 (109) | 22 (62) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 62 (97) | 52 (77) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 13 (19) | 19 (28) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 18 (19) | 11 (11) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 30 (43) | 29 (34) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 27 (38) | 19 (31) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 21 (27) | 15 (16) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 82 (128) | 78 (126) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 44 (55) | 48 (64) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 21 (22) | 18 (22) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 57 (98) | 61 (115) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 38 (60) | 27 (52) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 22 (27) | 26 (33) | 0 (0)
Dysgeusia (Nervous system disorders) | 15 (17) | 20 (24) | 0 (0)
Headache (Nervous system disorders) | 50 (76) | 57 (99) | 0 (0)
Migraine (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 81 (105) | 80 (97) | 0 (0)
Paraesthesia (Nervous system disorders) | 28 (38) | 26 (34) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 70 (81) | 78 (89) | 0 (0)
Anxiety (Psychiatric disorders) | 16 (16) | 13 (14) | 0 (0)
Insomnia (Psychiatric disorders) | 34 (35) | 27 (29) | 2 (2)
Dysuria (Renal and urinary disorders) | 22 (27) | 23 (29) | 0 (0)
Haematuria (Renal and urinary disorders) | 20 (25) | 15 (20) | 0 (0)
Incontinence (Renal and urinary disorders) | 3 (4) | 0 (0) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 5 (8) | 1 (1) | 2 (2)
Proteinuria (Renal and urinary disorders) | 54 (87) | 33 (52) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 16 (18) | 33 (39) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 17 (18) | 24 (26) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 25 (40) | 32 (40) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 40 (48) | 32 (41) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 (28) | 30 (34) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 31 (53) | 43 (65) | 1 (1)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 173 (173) | 179 (181) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 5 (8) | 6 (7) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 18 (18) | 9 (10) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 40 (58) | 26 (39) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 47 (66) | 36 (48) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 16 (20) | 9 (13) | 1 (2)
Hypertension (Vascular disorders) | 80 (117) | 71 (117) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT03635567/Prot_SAP_000.pdf